CLINICAL TRIAL: NCT04575116
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, CROSSOVER, SINGLE DOSE STUDY TO DETERMINE THE BIOEQUIVALENCE OF 12.2 MG TAFAMIDIS FREE ACID TABLET AND COMMERCIAL 20 MG TAFAMIDIS MEGLUMINE CAPSULE ADMINISTERED UNDER FASTED CONDITIONS TO HEALTHY PARTICIPANTS
Brief Title: A Study to Determine the Bioequivalence of Two Doses of Tafamidis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461095; Tafamidis (Other: Alias Study Number)
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tafamidis Free acid tablet then tafamidis meglumine capsule (Experimental): On Day 1 of each period, participants will receive a single dose of 1 of tafamidis formulations. Each period is separated by a washout of at least 16 days between administration of study drug.
  Interventions: Drug: Tafamidis free acid tablet; Drug: Tafamidis meglumine capsule
- Tafamidis meglumine capsule then Tafamidis Free acid tablet (Experimental): On Day 1 of each period, participants will receive a single dose of 1 of tafamidis formulations. Each period is separated by a washout of at least 16 days between administration of study drug.
  Interventions: Drug: Tafamidis free acid tablet; Drug: Tafamidis meglumine capsule

INTERVENTIONS:
Drug: Tafamidis free acid tablet — 12.2 mg tafamidis free acid tablet
Drug: Tafamidis meglumine capsule — 20 mg tafamidis meglumine soft gelatin capsule

SUMMARY:
Study to characterize the bioequivalence of a 12.2 mg free acid tablets compared to commercial supply (tafamidis meglumine soft gelatin 20 mg capsule) in healthy participants under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the ICD.
2. Healthy female participants of nonchildbearing potential and/or male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiovascular tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
4. BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
5. Capable of giving signed informed consent and compliance with study requirements and restrictions

Exclusion Criteria:

Medical Conditions:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb, or HCVAb. Hepatitis B vaccination is allowed.
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
5. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.

   Prior/Concurrent Clinical Study Experience:
6. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

   Diagnostic Assessments:
7. A positive urine drug test.
8. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
9. Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >450 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
10. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level greater than or equal to 1.5 × upper limit of normal (ULN);
    * Total bilirubin level greater than or equal 1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is greater than or equal ULN.

    Other Exclusions:
11. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
12. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
13. History of sensitivity to heparin or heparin induced thrombocytopenia.
14. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
15. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
16. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUCinf) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168
  Area under the plasma concentration time profile from time zero extrapolated to infinite time
Maximum observed plasma concentration (Cmax) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168
  Peak or maximum observed concentration

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC72) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72
  Area under the plasma concentration-time profile from time 0 to 72 hours post-dose
Area under the plasma concentration-time curve (AUClast) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168
  Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Mean residence time (MRT) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168
  Mean residence time (MRT)
Plasma Decay Half-Life (t1/2) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168
  Plasma Decay Half-Life (t1/2)
Number or percentage of patients with abnormal physical examination findings | Baseline up to Day 25
  Assessment of abnormal physical examination findings during study participation
Number or percentage of patients with change from baseline in Clinical Laboratory parameters | Baseline up to Day 25
  Change in clinical laboratory parameters
Number or percentage of patients with change from baseline in Vital sign measurements | Baseline up to Day 25
  Change in vital sign measurements
Number of patients with change in ECG parameters | Baseline up to Day 25
  Change in ECG parameters
Incidence of adverse events | Baseline up to Day 46
  Assessment of adverse events during study participation and up to 28 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461095